CLINICAL TRIAL: NCT02932644
Title: Association Between Baseline Vitamin D Metabolite Levels and Risk of Cardiovascular Events in Rheumatoid Arthritis Patients. A Cohort Study With Patient-record Evaluated Outcomes.
Brief Title: Vitamin D and Cardiovascular Events in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: The Danish Rheumatism Association (Other); University of Southern Denmark (Other); Region of Southern Denmark (Other); Pfizer (Industry); Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Mette Herly, MD, Odense University Hospital
Other Study IDs: 3-3013-930/1/
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Rheumatoid Arthritis; Cardiovascular Disease
Keywords: Rheumatoid Arthritis; Cardiovascular event; Cardiovascular mortality; Vitamin D
MeSH Terms: conditions — Arthritis, Rheumatoid; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis patients: Participants in the original, parental trial
  Interventions: Other: Baseline serum vitamin D level below 50 nmol/l; Other: Baseline serum vitamin D level at or above 50 nmol/l

INTERVENTIONS:
Other: Baseline serum vitamin D level below 50 nmol/l — There is no medical intervention. The two groups are simple allocated depending on serum levels of D-total at the time of diagnosis
Other: Baseline serum vitamin D level at or above 50 nmol/l — There is no medical intervention. The two groups are simple allocated depending on serum levels of D-total at the time of diagnosis

SUMMARY:
The aim of the study is to evaluate cardiovascular events during long-term follow-up in Rheumatoid Arthritis. The primary outcome "any cardiovascular event" will be evaluated using systematic audits of patient records, and will be associated to low levels of vitamin D at baseline, to investigate the hypothesis that low levels of vitamin D can be part of a prediction model for cardiovascular disease in Rheumatoid Arthritis.

DETAILED DESCRIPTION:
Cardiovascular morbidity and mortality is increased in patients with rheumatoid arthritis (RA), and among these patients, the prevalence of hypo-vitaminosis D is high. Low levels of vitamin D have been associated with elevated cardiovascular risk in healthy subjects. The objective of this study is to evaluate the risk of cardiovascular events in patients having low 25OHD-total levels at baseline compared to patients with sufficient levels, in an aggressively treated closed cohort of early-diagnosed RA patients.

The primary outcome will be the proportion of patients with any cardiovascular event, evaluated using systematic journal audits. Logistic regression models will be applied to test the hypothesis that there are more cardiovascular events in patients enrolled with a low level of vitamin D (< 50 nmol/l). Secondarily, Cox regression models, based on survival analysis, will be applied, to determine the extent to which independent variables (including different levels of vitamin D at baseline) predict not only whether a cardiovascular event occur, but also when it will occur.

ELIGIBILITY:
Inclusion Criteria: Fulfilling ACR1987 (American College of Rheumatology 1987 classification criteria for Rheumatoid Arthritis) criteria for RA, disease duration < 6 months, 2 or more swollen joints and age between 18 and 75 years -

Exclusion Criteria: Glucocorticoid treatment 4 weeks prior to inclusion, previous use of DMARDs, malignancy, diastolic blood pressure > 90 mm Hg, elevated serum creatinine, infections with parvovirus B19, Hepatitis B, C and HIV, and any condition contraindicating the study medication.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hundred-and-sixty early diagnosed and treatment-naive RA patients, recruited from five Danish University Clinics (Trial Centres) from October 1999 to October 2002
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 1999-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Cardiovascular event | Observed in the time-period from inclusion to October the 10th 2016
  Events will be recorded using systematic journal audits. A cardiovascular event will be further subclassified as shown in the secondary outcome measures, but for primary outcome measures; any cardiovascular event, including death, will serve as "an event"

SECONDARY OUTCOMES:
Acute cardiovascular hospitalisation due to Myocardial Ischamia | Observed in the time-period from inclusion to October the 10th 2016
  Non-fatal or fatal myocardial infarction, defined by National and International Guidelines (Thygesen et al. 1581-98).
  Fatal myocardial infarction is defined as primary fatal event within 7 days, documented post mortem by autopsy, or by the definition of myocardial infarction according to European Guidelines (Thygesen et al. 1581-98) Death of myocardial infarction as a consequence of medical examination/procedure/surgery will be classified as procedure related death.
  Acute Coronary Syndrome (ACS) includes acute ischaemic symptoms with eventual elevation in biomarkers or electrocardiographic changes which does not fulfil the criteria of acute myocardial infarction.
  Angina Pectoris. Revascularisation procedures (Percutaneous Coronary Intervention (PCI) or Coronary bypass Graft (CABG).
Acute cardiovascular hospitalisation due to hearth failure | Observed in the time-period from inclusion to October the 10th 2016
  Patients with non-elective hospitalisation or death, minimum one overnight stay, with symptoms or findings of heart failure.
  Death due to heart failure is defined as escalating heart failure symptoms prior to death.
Acute cardiovascular hospitalisation due to stroke | Observed in the time-period from inclusion to October the 10th 2016
  Cerebral haemorrhage, cerebral thromboembolism, Transitory Cerebral Ischemia (TCI) and others Stroke is defined as abrupt severe neurologic deficits, eventually with computer tomographic (CT) documentation. Death within 14 days after symptom-onset of stroke, and without other obviously reasons, is classified as caused by stroke
Acute cardiovascular hospitalisation due to arrhythmias | Observed in the time-period from inclusion to October the 10th 2016
  Atrial fibrillation or flutter, supraventricular tachycardia and others. Ventricular tachycardia, ventricular fibrillation and others. Death due to arrhythmia requires documentation, e.g. telemetric transcript, pacemaker or electrocardiogram
Acute cardiovascular hospitalisation due to Procedure-related cardiovascular event | Observed in the time-period from inclusion to October the 10th 2016
  Any cardiovascular event within 24 hours after cardiovascular medical examination/procedure/surgery.
Acute cardiovascular hospitalisation due to other reasons | Observed in the time-period from inclusion to October the 10th 2016
  Hospitalisation caused by other cardiovascular events, e.g. pulmonary embolism, rupture of aortic aneurism etc.
Acute cardiovascular hospitalisation due to supposed cardiovascular reason | Observed in the time-period from inclusion to October the 10th 2016
  Hospitalisation without any documented non-cardiovascular cause. All deaths which are not defined by the cardiovascular reasons mentioned above, and who are not caused by well-documented non-cardiovascular death.
  All deaths without known reason
Acute non-cardiovascular hospitalisation due to cancer | Observed in the time-period from inclusion to October the 10th 2016
  Acute hospitalisation due to cancer
Acute non-cardiovascular hospitalisation due to infection | Observed in the time-period from inclusion to October the 10th 2016
  Acute hospitalisation due to infection
Acute non-cardiovascular hospitalisation due to respiratory disease | Observed in the time-period from inclusion to October the 10th 2016
  Acute hospitalisation due to respiratory disease
Acute non-cardiovascular hospitalisation due to trauma | Observed in the time-period from inclusion to October the 10th 2016
  Acute hospitalisation due to trauma
Acute non-cardiovascular hospitalisation due to suicide | Observed in the time-period from inclusion to October the 10th 2016
  Acute - hospitalisation due to suicide
Acute non-cardiovascular hospitalisation due to other reasons | Observed in the time-period from inclusion to October the 10th 2016
  Acute hospitalisation du to other non-cardiovascular reasons, than those previous mentioned
Elective cardiovascular hospitalisation due to myocardial ischemia | Observed in the time-period from inclusion to October the 10th 2016
Elective cardiovascular hospitalisation due to arrhythmia | Observed in the time-period from inclusion to October the 10th 2016
Elective cardiovascular hospitalisation due to heart failure | Observed in the time-period from inclusion to October the 10th 2016
Elective cardiovascular hospitalisation due to other cardiovascular reasons | Observed in the time-period from inclusion to October the 10th 2016
Elective non-cardiovascular hospitalisation due to cancer | Observed in the time-period from inclusion to October the 10th 2016
Elective non-cardiovascular hospitalisation due to infection | Observed in the time-period from inclusion to October the 10th 2016
Elective non-cardiovascular hospitalisation due to respiratory disease | Observed in the time-period from inclusion to October the 10th 2016
Elective non-cardiovascular hospitalisation due to trauma | Observed in the time-period from inclusion to October the 10th 2016
Elective non-cardiovascular hospitalisation due to suicide | Observed in the time-period from inclusion to October the 10th 2016
Witnessed, sudden cardiovascular death | Observed in the time-period from inclusion to October the 10th 2016
  Death is witnessed and abrupt within one hour after symptom-onset
Non-witnessed, sudden cardiovascular death | Observed in the time-period from inclusion to October the 10th 2016
  Non-witnessed death with no obvious non-cardiovascular reasons (found death)
Non-sudden cardiovascular death | Observed in the time-period from inclusion to October the 10th 2016
  Death due to any of the cardiovascular caused previously mentioned, more than one hour after symptom-onset

CONTACTS AND LOCATIONS:
Overall Officials: Torkell Ellingsen, MD, Phd, Study Chair — Odense University Hospital

IPD SHARING:
Plan to Share IPD: Undecided